CLINICAL TRIAL: NCT01260467
Title: A Phase II Study of Memantine in the Treatment of Recurrent Glioblastoma
Brief Title: Memantine for Recurrent Glioblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Nimish Mohile, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RSRB34285; 054835-002 (Other Grant/Funding Number: American Society of Clinical Oncology)
Record Dates: First submitted 2010-12-10; First posted 2010-12-15 (Estimated); Results first posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-11

CONDITIONS: Glioblastoma
Keywords: recurrent
MeSH Terms: conditions — Glioblastoma; Recurrence | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- memantine arm (Experimental)
  Interventions: Drug: memantine

INTERVENTIONS:
Drug: memantine — 10 milligrams orally twice a day
  Other Names: Namenda

SUMMARY:
The purpose of this study is to determine if a medication called memantine is effective in treating glioblastoma. Memantine targets a specific receptor, called a glutamate receptor, which is thought to be involved in the growth of brain tumors. It has previously been studied for other types of conditions, such as Alzheimer's disease, but it has not yet been evaluated in the treatment of brain tumors. The investigators will also be determining how common it is for patients with brain tumors to have side effects to memantine. Memantine will be taken by mouth twice a day.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven World Health Organization (WHO) grade IV gliomas. Patients will be eligible if the original histology was a grade II or grade III glioma as long as a subsequent histological diagnosis of a grade IV glioma is confirmed.
* Patients must have shown unequivocal radiographic evidence for tumor progression by magnetic resonance imaging (MRI) scan. A scan should be performed within 10 days prior to registration and on a steroid dose that has been stable for at least 5 days. If the steroid dose is increased between the date of imaging and registration a new baseline MRI is required.
* Patients with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery (including gamma-knife or cyber-knife) must have confirmation of true progressive disease rather than radiation necrosis based upon either positron emission tomography (PET) or Thallium scanning, magnetic resonance spectroscopy (MRS), magnetic resonance perfusion, or surgical documentation of disease. The decision of which modality to use to make this confirmation will be at the discretion of the investigator.
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study. Patients must have signed an authorization for the release of their protected health information.
* Age greater than 18 years old, and with a life expectancy greater than 8 weeks.
* Karnofsky Performance Status greater or equal to 60
* Patients must have an interval of at least 28 days from any investigational agent or from prior cytotoxic therapy, 6 weeks from prior nitrosureas, 3 weeks from procarbazine and 2 weeks from vincristine.
* Patients must have failed prior radiotherapy and must have an interval of greater than 42 days from completion of initial radiation therapy to study entry or 28 days since radiation therapy used for recurrent tumor.
* Since memantine is not associated with myelosuppression, patients with persistent effects on bone marrow function from prior cytotoxic chemotherapies will be eligible as long as: white blood cells > 1,000/µl, absolute neutrophil count > 500/mm3, platelet count of > 50,000/mm3, and hemoglobin > 8 gm/dl). Patients must have adequate liver function and adequate renal function before starting therapy. These tests must be performed within 2 weeks prior to treatment initiation. Eligibility level for hemoglobin may be reached by transfusion.
* Patients must have a calculated creatinine clearance > 30 milliliters/minute.

Exclusion Criteria:

* Patients who are within 3 months of treatment with radiation and concurrent temozolomide will not be eligible unless there are new enhancing abnormalities outside the high dose radiation fields (i.e beyond the 80% isodose line) or surgical demonstration of active tumor.
* Patients must not be pregnant and must agree to practice adequate contraception. Women of childbearing potential must have a negative pregnancy test documented within 7 days prior to registration. Women must not be breastfeeding.
* Patients with a history of other cancer (except non-melanoma skin cancer or cancer of the cervix), unless in complete remission for at least 3 years are ineligible.
* Patients must not have any significant medical illnesses or other history that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy.
* Patients must not have any disease that will obscure toxicity or dangerously alter drug metabolism.
* Patients must not have prior or concurrent use of memantine or treatment with other N-methyl D-asparate (NMDA) receptor blocking therapies.
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of subject or legal guardian/representative to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nimish Mohile, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Agent Memantine Group: memantine:10 milligrams orally twice a day
Period: Overall Study
Arm/Group | Single Agent Memantine Group
Started | 4
Completed | 2
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Agent Memantine Group
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: 30 months
Population: not evaluated due to poor patient accrual
Arm/Group | Single Agent Memantine Group
Number analyzed (Participants) | 0

2. Primary Outcome: 6 Month Progression-free Survival
Time Frame: 24 months
Population: not evaluated due to poor patient accrual
Arm/Group | Memantine Arm
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Adverse Events
Description: This study will look at the number of participants who develop adverse events or side effects thought to be related to the memantine.
Time Frame: 24 months
Measure: Number; unit: participants
Groups:
- Single Arm: No adverse events reported.
Arm/Group | Single Arm
Number analyzed (Participants) | 4
participants | 0

ADVERSE EVENTS:
Groups:
- Single Agent Memantine Group: NO data to report
Arm/Group | Single Agent Memantine Group
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No